CLINICAL TRIAL: NCT04046965
Title: American Indian and Alaska Native Head Start Family and Child Experiences Survey (AIAN FACES 2019)
Acronym: AIAN FACES
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 50515B
Record Dates: First submitted 2019-05-28; First posted 2019-08-06 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Head Start Participation
Keywords: Alaska natives; child care; child development; child health; child rearing; children; curriculum; early childhood education; families; Head Start; Native Americans; parenting skills; parents; programs; school readiness; teachers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Region XI Head Start children and families - Fall 2019 to Spring 2020: children (720) parents (720) classrooms/teachers (85) program directors (22) center directors (40)

SUMMARY:
The American Indian and Alaska Native Head Start Family and Child Experiences Survey (AIAN FACES) 2019 builds on AIAN FACES 2015 (NCT03842111), which was the first national study children and families participating in Region XI Head Start. In consultation with the AIAN FACES Workgroup, Mathematica developed instruments and data collection procedures to assess the school readiness skills of 720 children and survey their parents and Region XI Head Start teachers in fall 2019 and spring 2020; conduct observations in those children's Region XI Head Start classrooms; and survey Region XI Head Start staff in spring 2020. Due to the COVID-19 pandemic, spring 2020 child assessments and classroom observations were canceled after two weeks, while surveys of parents and staff continued.

DETAILED DESCRIPTION:
The design and execution of AIAN FACES has been informed by close collaboration with members of the AIAN FACES Workgroup which includes Region XI Head Start program directors, researchers with experience working with AIAN communities, Mathematica study staff, and federal officials from the Office of Head Start and the Office of Planning, Research and Evaluation.

Building on AIAN FACES 2015 as the foundation, members of the AIAN FACES Workgroup have shared insights and information on the kinds of information needed about children and families served by Region XI AIAN Head Start programs. Members also provided input on recruitment practices and study methods that are responsive to the unique cultural and self-governing contexts of tribal Head Start programs. They also consulted on priorities for dissemination and drafts of dissemination products.

AIAN FACES 2019 provides the mechanism for collecting data on a nationally representative probability sample in Region XI to provide valid and reliable information to federal, local, and tribal community stakeholders. AIAN FACES 2019 focuses on children and families to describe the school readiness skills, family characteristics, and Head Start experiences of these children, with a focus on Native culture and language. The investigators collected information on programs and classrooms to provide context for children's experiences. Data collection with Region XI children, families, classrooms, and programs took place in the Fall of 2019 and the Spring of 2020. Originally, AIAN FACES 2019 also sought to describe classroom quality for children in Region XI, but was unable to do so, with classroom observations cancelled after two weeks due to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria: the Region XI Head Start programs participating in AIAN FACES 2019 were a probability sample selected from among 146 study-eligible programs on the 2017-2018 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be:

* Providing services directly to children ages 3 to 5
* The Head Start Program Performance Standards require that children turn 3 by date used to determine eligibility for public school in the community in which the Head Start program is located. Therefore, some study children were 2 years old at the time of sampling if sampling occurred before the date used for public school eligibility.
* Not be in imminent danger of losing its grantee status. Probability samples of centers were selected within each program, classrooms within each center (within those classrooms, eligible classrooms needed to have at least one Head Start child enrolled) and children within each classroom. Teachers associated with selected classrooms were included in the study with certainty, as were parents associated with selected children.

Exclusion Criteria: Head Start programs in Regions I through X and Migrant and Seasonal Head Start (Region XII) were not eligible for AIAN FACES. Other ACF studies (FACES-NCT03971435 and MSHS-NCT03116243) focus on those programs.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Region XI Head Start children (and their families), Region XI Head Start programs, Region XI Head Start centers, Region XI Head Start classrooms/teachers
Sampling Method: Probability Sample
Enrollment: 1587 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
English proficiency | October to December 2019, March 2020
  Children's English language proficiency were assessed during week-long site visits using Preschool Language Assessment Survey (preLAS 2000): Simon Says and Art Show. See Duncan and DeAvila for more information on the scores and technical properties.
Language-English receptive vocabulary | October to December 2019, March 2020
  Indicators of language were assessed during week-long site visits using Peabody Picture Vocabulary Test-Fifth Edition (PPVT-5). See Dunn 2019 for more information on the scores and technical properties.
  Dunn, D. M. Peabody Picture Vocabulary Test, Fifth Edition. Examiner's Manual and Norms Booklet. Bloomington, MN: NCS Pearson, Inc., 2019.
Language-Expressive vocabulary | October to December 2019, March 2020
  Indicators of language were assessed during week-long site visits using Expressive One-Word Picture Vocabulary Test-Fourth Edition (EOWPVT-4 or EOWPVT-4 Spanish-Bilingual Edition). See Martin and Brownell 2010 and Martin 2012 for more information on the scores and technical properties.
Literacy-Letter word knowledge | October to December 2019, March 2020
  Indicators of literacy were assessed during week-long site visits using Letter-Word Identification Test from Woodcock-Johnson IV Tests of Achievement-Fourth Edition. Please see Schrank et al. 2014 and Woodcock et al. 2004 for more information on the scores and technical properties.
Literacy-early writing | October to December 2019, March 2020
  Indicators of literacy were assessed during week-long site visits using Spelling Test from Woodcock-Johnson IV Tests of Achievement-Fourth Edition. Please see Schrank et al. 2014 and Woodcock et al. 2004 for more information on the scores and technical properties.
Literacy-Letter sounds knowledge | October to December 2019, March 2020
  Indicators of literacy were assessed during week-long site visits using ECLS-B Letter Sounds. Please see Snow et al. 2007 for more information on the scores and technical properties Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. "Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06)." NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
Mathematics | October to December 2019, March 2020
  Indicators of mathematics were assessed during week-long site visits using the Early Childhood Longitudinal Study-Birth Cohort (ECLS-B) preschool mathematics assessment of children's understanding of relative size, ordinal numbers, and pattern matching; number recognition; and the children's ability to count, recognize shapes, add, and solve word problems. Please see Snow et al. 2007 for more information on the scores and technical properties.
Mathematics | October to December 2019, March 2020
  Indicators of mathematics were assessed during week-long site visits using the Woodcock-Johnson IV Tests of Achievement-Fourth Edition (Applied Problems Test). Please see Schrank et al. 2014 for more information on the scores and technical properties.
Children's physical health | October to December 2019, March 2020
  Indicators of physical well-being were assessed by weighing (using kilograms) and measuring children's height (using centimeters), and combining these measurements to calculate Body Mass Index (BMI) in in kg/m^2.
General health status | October to December 2019, March 2020
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor
Executive function | October to December 2019, March 2020
  Indicators of executive function were assessed by the Minnesota Executive Function Scale (MEFS). The MEFS is a standardized and adaptive assessment administered on a touch-screen tablet with child-friendly graphics, avatars, and child-directed instructions. The MEFS provides an objective assessment of children's self-regulation, particularly cognitive flexibility, working memory, and inhibitory control. See Carlson and Zelazo for more information.
Social-emotional development | October-December 2019, March-July 2020
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the AIAN FACES 2019 User's Manual (Bernstein et al. 2021a) for more information on the scores and technical information.
Social-emotional development-cognitive/social behaviors | October-December 2019, March-July 2020
  Indicators of social-emotional development were assessed using assessor report children's cognitive/social behaviors during the assessment time, using the Leiter International Performance Scale-Third Edition Examiner Rating Scale. The Leiter comprises eight subscales that examine children's approach to the assessments, their engagement with the materials, and their ability to attend to and regulate their physical and emotional responses during the assessment tasks. Please see Roid et al. 2013 for more information on the scores and technical properties.
Social-emotional development - Approaches to learning | October-December 2019, March-July 2020
  Indicators of social-emotional development were assessed using teacher report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
Classroom quality-teacher child interactions | One-day observation in March 2020
  Indicators of classroom quality were assessed using the the PreK Classroom Assessment Scoring System. The Pre-K CLASS assesses the qualities of interactions between teachers and students in classrooms and measures aspects of interactions related to children's early academic achievement and social competencies. Please see Pianta et al. 2008 for more information on the scores and technical properties.
Classroom quality-global classroom environment | One-day observation in March 2020
  Indicators of classroom quality were assessed using a shortened form of the Early Childhood Environment Rating Scale-Revised (ECERS-R), a global rating of classroom quality based on structural features of the classroom (Harms et al. 2005). The items in the short form represent the strongest 21 items identified by researchers in a large-scale study (Clifford et al. 2005). Please see Harms et al. 2005 and Clifford et al. 2005 for more information on the scores and measure technical properties.
Classroom quality-Native cultural and language classroom observation | One-day observation in March 2020
  In AIAN FACES 2019, children's exposure to Native cultural and language experiences during the classroom observation were documented using the Native Culture & Language in the Classroom Observation (NCLCO). The NCLCO was developed for AIAN FACES 2015 and adapted for 2019, both with the guidance of the study Workgroup. Please see AIAN FACES 2019 Workgroup 2021 for more information.
Parents' depressive symptoms | October-December 2019, March-July 2020
  Parents' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Teachers' depressive symptoms | October-December 2019, March-July 2020
  Teachers' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bernstein, Ph.D., Study Director — Mathematica Policy Research; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research
Locations (1):
- Mathematica Policy Research, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In the future, AIAN FACES 2019 archived data will be available for access.
Time Frame: Data from 2019 and 2020 are currently available.
Access Criteria: Access to AIAN FACES 2019 data is limited to individuals working in institutions of higher education or research organizations. In addition to completing the Inter-university Consortium for Political and Social Research (ICPSR) standard application, researchers must complete additional requirements in order to obtain access to the AIAN FACES 2019 data.

REFERENCES:
- [Background] Bernstein, S., A. Kopack Klein, B. Lepidus Carlson, A. Li., N. Aikens, M. Dang, M. Scott, S. Skidmore, M. Cavanaugh, J. Cannon, and contributing authors. "American Indian and Alaska Native Head Start Family and Child Experiences Survey 2019: User's Manual." Report submitted to the Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services, Washington, DC: Mathematica, 2021.
- [Background] Carlson, S. M., & Zelazo, P. D. (2014). Minnesota Executive Function Scale: Test Manual. Reflection Sciences, Inc. St. Paul, MN.
- [Background] Clifford, Richard, Oscar Barbarin, Florence Chang, Diane M. Early, Donna Bryant, Carollee Howes, Margaret Burchinal, and Robert Pianta. What Is Pre-Kindergarten? Characteristics of Public Pre-Kindergarten Programs. Applied Developmental Science, vol. 9, no. 3, 2005, pp. 126-143.
- [Background] Duncan, S.E., and E. DeAvila. Preschool Language Assessment Survey 2000 Examiner's Manual: English Forms C and D. Monterey, CA: CTB/McGraw-Hill, 1998.
- [Background] Dunn, D. M. Peabody Picture Vocabulary Test, Fifth Edition. Manual. Bloomington, MN: NCS Pearson, Inc., 2019.
- [Background] Harms, T., R.M. Clifford, and D. Cryer. Early Childhood Environment Rating Scale: Revised Edition. New York. Teachers College Press, 2005.
- [Background] EOWPVT-4: Martin, N., and R. Brownell. "Expressive One-Word Picture Vocabulary Test-4th Edition." Novato, CA: Academic Therapy Publications, 2010.
- [Background] Pianta, Robert, K. LaParo, and B. Hamre. The Classroom Assessment Scoring System Pre-K Manual. Charlottesville, VA: University of Virginia, 2008.
- [Background] Radloff, L. "The CES-D Scale: A Self-Report Depression Scale for Research in the General Population." Applied Psychological Measurement, vol. 1, no. 3, 1977, pp. 385-401.
- [Background] Roid, G.H., L.J. Miller, M. Pomplu, and C. Koch. Leiter International Performance Scale-3rd Edition. Wood Dale, IL: Stoelting, 2013.
- [Background] Schrank, F., K. McGrew, and N. Mather. Woodcock-Johnson IV. Rolling Meadows, IL: Riverside, 2014.
- [Background] Snow, K., L. Thalji, A. Derecho, S. Wheeless, J. Lennon, S. Kinsey, J. Rogers, M. Raspa, and J. Park. Early Childhood Longitudinal Study, Birth Cohort (ECLS-B), Preschool Year Data File User's Manual (2005-06). NCES 2008-024. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2007.
- [Background] U.S. Department of Education, National Center for Education Statistics. Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade. NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.
- See also: To learn more about AIAN FACES and access reports/publications, please visit the AIAN FACES ACF website. — https://www.acf.hhs.gov/opre/project/american-indian-and-alaska-native-head-start-family-and-child-experiences-survey-ai-0
- See also: To learn more about AIAN FACES and access reports/products, individuals may also visit the Mathematica study website. — https://mathematica.org/projects/american-indian-and-alaska-native-head-start-family-and-child-experiences-survey-ai-an-faces